CLINICAL TRIAL: NCT04175821
Title: Dept. of Radiation Oncology, PGIMER, Chandigarh
Brief Title: Late-term Effects of Hypofractionated Chest Wall and Regional Nodal Irradiation in Patients With Breast Cancer
Acronym: LEHR
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: LEHR
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Late Effects of Hypofractionated Radiotherapy in Breast Cancer
Keywords: Breast cancer; Hypofractionated radiotherapy; Post mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 35Gy/ 15#/3weeks to chest wall and 40Gy/15#/3 weeks to supraclavicular fossa

SUMMARY:
Survival of breast cancer patients has improved with multimodality treatment. Hypofractionated radiotherapy (RT) is rapidly emerging as one of the options for breast cancer patients after breast conservation surgery (BCS) but data on postmastectomy radiation therapy (PMRT) with hypofractionation is lacking and there is always concern for the late effects of RT especially with regional nodal irradiation (RNI). The potential survival benefits of locoregional radiation needs to be balanced with late-term effects. There is a dearth of data on RNI with hypofractionation. Therefore, reporting late-term effects of radiation in these patients is of utmost importance, especially with hypofractionation. Very few patients were given PMRT or RNI in the START trials, so definitive conclusions about the safety of shorter fractionation RNI cannot be drawn from these studies.1-3 There are also studies from Canada and the US with similar dose fractionations in the PMRT setting with limited number of patients but without RNI.4,5 There is a world-wide need for data on PMRT and especially with RNI for patients with breast cancer with its late-term consequences. Because of this, many radiation oncology societies are hesitant in recommending hypofractionated RNI. It is also an area for potential research in breast cancer radiotherapy. We have published our clinical outcomes with 3 weeks of adjuvant local and RNI with hypofractionation in the past.6-10 In this study, we will report late-term effects of PMRT and RNI with this schedule in patients with stage II and III breast cancer from a single institute from India which is practicing hypofractionation since 1976.

DETAILED DESCRIPTION:
Between January 1990 to December 2007, women with breast cancer who were given radical treatment with mastectomy, systemic therapy and RT at least 10 years ago were included. Eligible patients were recruited from the radiotherapy department record and these were on regular follow-up in the breast clinic. The study was approved by the departmental ethics committee. Clinical, pathological and treatment characteristics were taken from the patient file. Inclusion criteria were: female patients age ≥18 years of age, with invasive carcinoma of the breast, post mastectomy, complete microscopic excision of primary tumour and stage II or III disease treated with locoregional RT. Exclusion criteria were: breast conserving surgery, stage I or IV disease, past history of malignancy except (i) basal cell skin cancer or CIN cervix uteri or(ii) non-breast malignancy if treated with curative intent and at least 5 years disease-free or contralateral breast cancer, including ductal carcinoma in situ (DCIS), irrespective of date of diagnosis. Patients with bilateral breast cancer were also excluded.

Patients were treated in supine position on a breast board with ipsilateral arm abducted to 900. All patients were planned using 2-D fluoroscopic conventional simulator with two tangential fields to the chest wall and a single incident field to the axilla and supraclavicular fossa. Lateral border of supraclavicular fossa was up to deltoid insertion.

Radiotherapy dose delivered was 35Gy/15fractions /3 weeks to the chest wall. Dose was prescribed at mid separation. Bolus was used in all patients on alternate days, that is for 50% of treatment. In patients with positive margins bolus was used daily and a scar boost of 10Gy/4fractions was given. None of the patients had breast reconstruction. Supraclavicular fossa(SCF), axillary chain and internal mammary nodal irradiation (IMNI)6 was done with a single incident field. No posterior axillary field was used. The dose delivered was 40Gy/15fractions/3weeks. All patients were treated on linac or cobalt-60 machine.

A biologically effective dose(BED) of 35Gy/15fractions/3weeks is 75.1Gy in terms of 2Gy per fraction for late effects, 55.1Gy for tumour control, 45Gy for erythema and 42.3Gy for desquamation in case of local radiotherapy. The BED for RNI with this schedule is 90Gy, 65Gy, 52.5Gy and 49Gy for late effects, tumour control, erythema and desquamation, respectively.

Patients were seen by the radiation oncologists with special focus on chest wall fibrosis, telangiectasia, shoulder function, lymphedema, arm pain and sensory symptoms. Late fibrosis was defined grade 1 as barely palpable firmness, grade 2 as definite increased firmness and grade 3 as marked firmness of the chest wall. Telangiectasia was defined grade 1 as <1cm2, grade 2 as 1 cm2-4 cm2 and grade 3 as >4 cm2 area of chest wall. Lymphedema was graded by measuring arm circumference 10cm above and below the medial epicondyle of humerus . For lymphedema and shoulder function, the treated side was compared with the untreated opposite side as a reference. Lymphedema was classified as none, mild, moderate and marked if there was no difference, 0.5-2cm, 2.1-3cm and >3cm difference, respectively in the circumference of the affected and normal arm. If the patient had symptoms of pain in the arm, paresthesia, numbness, weakness, or other sensory symptoms then injury to the brachial plexus was suspected and reported as brachial plexopathy. A four point scale(none, a little, quite a bit, very much ) was used to assess all late effects according to the RTOG LENT SOMA scale. Late lung toxicity was defined grade 1 as asymptomatic or mild symptoms of dry cough, slight radiographic changes; grade 2 as moderate symptomatic fibrosis or pneumonitis (severe cough), low grade fever, patchy radiographic changes; grade 3 as severe symptomatic fibrosis or pneumonitis, dense radiographic changes and grade 4 as severe respiratory insufficiencies, oxygen required of assisted ventilation. Late cardiac toxicity was defined grade 1 as minimal enlargement of cardiosilhoutte (ECS), grade 2 as ECS without pulmonary congestion, grade 3 as ECS pulmonary congestion and grade 4 as ECS with frank pulmonary oedema. All late effects assessment scores were dichotomised as none/mild versus moderate/marked effects.

ELIGIBILITY:
Inclusion Criteria:

* invasive carcinoma of the breast, post mastectomy complete microscopic excision of primary tumour and stage II or III disease

Exclusion Criteria:

* breast conserving surgery, stage I or IV disease, past history of malignancy except (i) basal cell skin cancer or CIN cervix uteri or(ii) non- breast malignancy if treated with curative intent and at least 5 years disease-free or contralateral breast cancer, ductal carcinoma in situ (DCIS), bilateral breast cancer

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who had undergone mastectomy followed by radiotherapy to the chest wall and regional nodes. Chemotherapy and hormonal therapy depending on the indication.
Sampling Method: Non-Probability Sample
Enrollment: 1770 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2007-12-31 (Actual); Study Completion 2019-06

PRIMARY OUTCOMES:
Chest wall fibrosis ("change" is being assessed) | 5, 10 and 15 years
  Late fibrosis was defined grade 1 as barely palpable firmness, grade 2 as definite increased firmness and grade 3 as marked firmness of the chest wall.

SECONDARY OUTCOMES:
Telengiectasia ("change" is being assessed for all outcomes) | 5, 10 and 15 years
  Telangiectasia was defined grade 1 as <1cm2, grade 2 as 1 cm2-4 cm2 and grade 3 as >4 cm2 area of chest wall
Lymphedema | 5, 10 and 15 years
  Lymphedema was graded by measuring arm circumference 10cm above and below the medial epicondyle of humerus . For lymphedema and shoulder function, the treated side was compared with the untreated opposite side as a reference. Lymphedema was classified as none, mild, moderate and marked if there was no difference, 0.5-2cm, 2.1-3cm and >3cm difference, respectively in the circumference of the affected and normal arm.
Lung toxicity | 5, 10 and 15 years
  Late lung toxicity was defined grade 1 as asymptomatic or mild symptoms of dry cough,slight radiographic changes; grade 2 as moderate symptomatic fibrosis or pneumonitis (severe cough), low grade fever, patchy radiographic changes; grade 3 as severe symptomatic fibrosis or pneumonitis, dense radiographic changes and grade 4 as severe respiratory insufficiencies, oxygen required of assisted ventilation.
Cardiac toxicity | 5, 10 and 15 years
  Late cardiac toxicity was defined grade 1 as minimal enlargement of cardiosilhoutte (ECS), grade 2 as ECS without pulmonary congestion, grade 3 as ECS pulmonary congestion and grade 4 as ECS with frank pulmonary oedema. All late effects assessment scores were dichotomised as none/mild versus moderate/marked effects.